CLINICAL TRIAL: NCT00226798
Title: Interleukin-2, Interferon Alpha,Capecitabine and Vinblastin for Treatment of Metastatic Renal Cell Carcinoma: A Multicenter Study
Brief Title: Immunochemotherapy for Metastatic Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Roche Pharma AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1747CTIL; Raphael Rubinov
Record Dates: First submitted 2005-09-26; First posted 2005-09-27 (Estimated); Last update posted 2006-01-04 (Estimated); Status verified 2005-09

CONDITIONS: Adenocarcinoma Clear Cell
MeSH Terms: conditions — Adenocarcinoma, Clear Cell | interventions — Capecitabine

INTERVENTIONS:
Drug: Capecitabine (Xeloda)

SUMMARY:
Immunochemotherapy consisting of IL-2, INF-A, and VBL and 5FU is regarded as the treatment of choice in metastatic renal cell carcinoma. During the period 1996-2000, we evaluated the efficacy and toxicity of this immunochemotherapy, combined with an aggressive surgical approach: nephrectomy before treatment and resection of residual disease. The 3-year survival rate for the entire group and complete responder patients was 30% and 88%, respectively. The side effects were usually moderate and consisted mainly of a flu-like syndrome, headache, nausea, vomiting and depression. Most importantly, there was no drug-related death. Good performance status, absence of bone metastases and prior nephrectomy were associated with higher response rates.

Capecitabine is a novel fluoropyrimidine carbamate, orally administered and selectively activated to Fluorouracil by a sequential triple-enzyme pathway in liver and tumor cells. Capecitabine at dose of 2,500mg/m2/d divided equally into two daily doses for 14 days in patients who failed to respond to "standard" immunotherapy achieved a 30% objective response. Toxicity consisted of hand-foot syndrome.

Aim of Study:

To evaluate efficacy and toxicity of the combination of IL-2, INF-A, VBL and Capecitabine in MRCC

DETAILED DESCRIPTION:
This is a phase II study, non-randomized in patients with metastatic renal cell carcinoma. The treatment will include: Proleukin (produced by Chiron and supplied by Megapharm Israel Ltd), Roferon A and Xeloda (produced by Roche) and VBL. The treatment will be given in 8-week courses with an interval of two weeks of rest in which the response (on D63) and toxicity will be assessed.

45 patients with MRCC will be entered into this study during a 18-month period. All patients must meet all inclusion and exclusion criteria. All data of each participating patient, including medical history, disease characteristics, laboratory and imaging tests, response and toxicity to treatment will be entered into the specific form before, during, after each treatment course and during follow up.

Patients will be followed up for survival status and disease status every 6 months until last visit or death.

Treatment Schedule:

Proleukin S.C. 10X106 IU/m2 three times a week (Sun, Tue, Thu), weeks 1 - 4 Roferon A S.C. 6 X 106 IU/m2 once a week (Wed), weeks 1 - 4 Roferon A S.C. 3 X 106 IU/m2 three times a week, weeks 5 - 8 Xeloda Oral 1,000 mg/m2 twice a day, weeks 5, 6 Vinblastine I.V. 4mg/m2, Day 1, weeks 5 &

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria; Patients with the following criteria will be included in this study

* Pathological (histology or cytology) diagnosis of renal cell carcinoma
* Clinical evidence of metastatic disease
* Performance status 0 - 2 (European Cooperative Oncology Group Score)
* Nephrectomy before starting treatment
* Normal cardiac function (left ventricular ejection fraction >45%).
* Normal blood counts: WBC >3,000/ml3, Hb >10gr%, Platelets >100,000/ml3
* Normal kidney function: Creatinine <1.3 mg/dl
* Age  18 years
* Patient's written consent (on informed consent form)

Exclusion Criteria:

* Life expectancy less than 3 months
* Brain metastases
* Ischemic heart disease - active
* Prior immunochemotherapy
* Performance status 3 or more (European Cooperative Oncology Group Score)
* Schizophrenia
* Active liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2003-12; Study Completion 2005-09

PRIMARY OUTCOMES:
Objective response

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Eliahu Gez, MD, Study Chair — Rambam Health Care Campus
Locations (1):
- Rambam medical Center, Haifa, Israel